CLINICAL TRIAL: NCT04927949
Title: Evaluation of Myocardial Reperfusion and Residual Thrombotic Burden After Primary PCI for STEMI in Patients With High on Ticagrelor Platelet Reactivity Treated by IV Cangrelor Versus Ticagrelor Alone
Brief Title: Evaluation of Myocardial Reperfusion After Primary PCI in Patients With High Platelet Reactivity Treated by Cangrelor or Not
Acronym: ERMIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-126
Record Dates: First submitted 2021-05-27; First posted 2021-06-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-01

CONDITIONS: ST-elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- patients without HPR (Sham Comparator): standard primary PCI
  Interventions: Procedure: standard PCI
- patients with HPR randomized to cangrelor (Experimental): Cangrelor perfusion started before PCI
  Interventions: Drug: cangrelor perfusion during PCI
- patients with HPR randomized to standard of care (Placebo Comparator): standard primary PCI
  Interventions: Procedure: standard PCI

INTERVENTIONS:
Drug: cangrelor perfusion during PCI — Cangrelor perfusion (started before PCI) with intravenous bolus of 30 microgram/kg, followed by a perfusion of 4 microgram/kg/min during 2 hours or until the end of the PCI if longer
  Arms: patients with HPR randomized to cangrelor
Procedure: standard PCI — primary PCI without cangrelor
  Arms: patients with HPR randomized to standard of care; patients without HPR

SUMMARY:
This study aims to evaluate the impact on myocardial reperfusion and residual thrombotic burden of adding Cangrelor -a potent and immediate P2Y12 inhibitor- to ticagrelor in primary PCI patients with high on ticagrelor platelet reactivity compared to standard of care with ticagrelor alone.

DETAILED DESCRIPTION:
Despite the use of potent P2Y12 inhibitor such as ticagrelor, half of the patients presented high platelet reactivity (HPR) at the time of primary percutaneous coronary intervention (PCI) for ST-elevation myocardial infarction (STEMI). HPR has been associated with impaired myocardial reperfusion. Myocardial reperfusion, assessed using myocardial blush grade, is a strong prognostic factor associated with infarct size and mortality. Antiplatelet therapy intensification using a potent and immediate P2Y12 inhibitor such as Cangrelor according a point-of-care platelet function test has not been studied in the acute phase of STEMI.

This study aims to evaluate the impact on myocardial reperfusion and residual thrombotic burden of adding Cangrelor to ticagrelor in primary PCI patients with high on ticagrelor platelet reactivity compared to standard of care with ticagrelor alone.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted for STEMI within 24 hours from symptom onset
* pretreated with ticagrelor, aspirin and enoxaparin (according local protocol)
* successfully treated by primary PCI of a native coronary culprit lesion
* anatomy accessible to optical coherence tomography (OCT or OFDI)

Exclusion Criteria:

* cardiogenic shock
* stent restenosis or thrombosis
* use of glycoprotein IIb/IIIa inhibitors before or during PCI
* known coagulation disease
* high bleeding risk (thrombocytopenia <100,000/dL, surgery <30 days, active bleeding)
* uncontrolled arterial hypertension (>180/110 mmHg)
* history of stroke (ischemic or hemorrhagic) or transient ischemic attack
* known severe renal insufficiency (eGFR <30 ml/min)
* oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Grade of myocardial blush | during procedure
  myocardial blush grade from 0 to 3 (normal)

SECONDARY OUTCOMES:
percentage of residual thrombus burden | during procedure
  intrastent residual thrombus burden assessed by optical coherence tomography
measure of platelet reactivity | during procedure
  Platelet reactivity using VerifyNow after PCI for patients with basal platelet reaction unit>208
troponin | day 1
  peak value
infarct size and no reflow on MRI | during hospitalization assessed up to 7 days
clinical outcomes | during hospitalization assessed up to 7 days
  death, new myocardial infarction, stent thrombosis, new revascularization, stroke, major bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France